CLINICAL TRIAL: NCT04821804
Title: Local Application of Hyaluronic Acid (HYADENT BG) With Free Soft Tissue Grafing Improves Treatment Outcomes.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JordanUST6
Record Dates: First submitted 2020-10-11; First posted 2021-03-30 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Gingival Recession, Plastic Surgery
Keywords: tooth, gingiva, soft tissue graft
MeSH Terms: conditions — Gingival Recession | interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): local application of HYADENT BG on both donor and recipient sites
  Interventions: Drug: Hyaluronic Acid (HYADENT BG)
- control (Placebo Comparator): application of normal saline on both donor and recipient sites
  Interventions: Drug: Hyaluronic Acid (HYADENT BG)

INTERVENTIONS:
Drug: Hyaluronic Acid (HYADENT BG) — the operator topically applied the HYADENT BG on the borders of the graft after stabilization.
  on the donor site and injection of HYADENT BG in collagen sponge that was placed over the site, then figure X sutures to close the area using (4-0 polyglycolic acid/ reverse cutting/ 12 mm) resorbable sutures

SUMMARY:
A total of 24 healthy non-smoker patients requiring FGG recruited for the study. Subjects were equally and randomly assigned into two groups. Test group, local application of HYADENT BG on both donor and recipient sites. Control group, application of normal saline on both sites as placebo. The FGG dimensions were evaluated at 1, 3- and 6-month recall using digital photographs. Post-operative pain was evaluated for 14 days. Color matching and patient satisfaction were evaluated at 6 months.

DETAILED DESCRIPTION:
The study was approved in the Institutional Review Board (IRB) at Jordan University for Science and Technology and Jordanian Food and Drug Administration. This clinical trial was a single-centre, parallel-group, prospective, randomized, subject-blind placebo-controlled study of Hyaluronic Acid (HYADENT BG), and placebo in patients undergoing FGG who met the inclusion criteria. The study was performed in accordance with the International Conference on Harmonization Good Clinical Practice and CONSORT guidelines.For all patients included in the study, phase I periodontal therapy was completed 4 weeks pre-surgically. All Patients were instructed to gargle with anti-microbial chlorohexidine mouth 0.2% for one minute pre-surgically to eliminate any source of infection. local anesthesia injection by 2% lidocaine with 1:100 000 epinephrine was given into the depth of the vestibule.

On the recipient site, coronal incision was made horizontally at the level of MGJ on the teeth to be treated and passing the midpoint of the adjacent teeth, at right angle 90 degree to the Mesio-angle and Disto-angle to the papilla to create "Butt joint" margin. The recipient sites had even thickness of the flap, then the flap was repositioned apically On the palatal donor site, custom tinfoil template was placed over the palatal mucosa to outline the dimensions of the graft according to the recipient bed. The area that chosen to harvest the graft was between first premolar and first molar and located 2 mm distant from the gingival margins of the corresponding teeth. After harvesting the FGG, Photograph was taken immediately to measure the graft area at the baseline. Connective tissue surface was carefully inspected for irregularities or adipose tissue after graft separation to minimize dead space between the graft and the recipient bed and enable quick revascularization of the graft. Graft thickness was immediately confirmed with a digital caliber at 5 points (four corners and center of the graft) and, if necessary, the graft was prepared (thinned) while holding it on sterile tongue depressor to obtain a graft approximately 1 to 1.3 mm thick.

For donor site closure, in the test group, application of HYADENT BG on the donor site and injection of HYADENT BG in collagen sponge that was placed over the site, then figure X sutures to close the area using (4-0 polyglycolic acid/ reverse cutting/ 12 mm) resorbable sutures. On the other hand, control group donor sites were washed with normal saline and placing the collagen sponge that soaked in normal Saline on the donor site. For both donor tested and control sites, a collagen sponge and figure X -0 resorbable sutures were placed. Finally, covering the donor areas in both groups with Septo-pack gingival dressing (Septodont, Saint Maur-des-fosses, France) then X suture over the pack to prevent the displacement of pack (Figure 1a,b).

For the graft stabilization, in the study group, application of HYADENT BG on the surgical site and the borders also was established. On the other hand, control group recipient bed was washed with normal saline before the graft placement. Minimal and fixed number of sutures was used for stabilization of the FGG as described previously by (Sullivan, 1968). 11 Magnification using Dental magnification loupe (3.5X- 420mm) was used to obtain the graft stabilization by sutures. Graft stabilized in both groups using (6-0 polyglycolic acid/ reverse cutting/ 12 mm suture) with two simple interrupted sutures in the coronal portion of the two Apico-coronal edges, and one suture in the mid-point of the coronal border using simple interrupted method. One Periosteal Oschenbein suture (4-0 polyglycolic acid/ reverse cutting/ 12 mm suture) to fix the graft on its place. In the study group, the operator topically applied the HYADENT BG on the borders of the graft after stabilization. On the other hand, in control group, operator topically applied normal saline on the bed before stabilization of the graft as placebo. Finally, after stabilization, gentle pressure was applied to the graft for five minutes in both groups to stabilize the clot under the graft

Clinical photographs Clinical photographs were used to measure the surface area of the graft in all follow up periods, and to assess the color matching between the grafted area and the adjacent tissue at the end of the final follow-up visit on 6-month period. All intra oral photographs were taken with the same professional camera (Nikon D3400) with same intraoral photographs setting (Aperture 32, Shutter speed 1/160, ISO 100), professional macro lens (Sigma 105mm f/2.8 EX DG OS HSM Macro Lens), ring flash (Godox Macro Ring Flash ML-150) with ½ light exposure. Fixed distance between the chin of the patient and the ring flash was considered to take the photograph was 30 cm. Lip retractor was used to allow uniform lighting of the area, and using Michigan "O" periodontal probe parallel with adjacent teeth as a reference (known distance between two fixed points) for measuring the graft area using the digital software.

Postoperative protocol The post-operative care aimed at maintaining wound stability. Post-operative instructions included ceasing tooth brushing and flossing around the surgical sites until the day of periodontal sutures removal (day 14). However, Patients were directed to start brushing their teeth expect the experimental area (canine to canine) after one week and to eat only soft foods during the first week and to avoid any mechanical or thermal trauma. No antibiotics nor analgesics were prescribed. Patients were followed professionally by the same periodontist (S.K), scheduled to be seen on month 1, 3, and 6 months.

Parameters Visual analogue scale (VAS) was used to evaluate the pain for two weeks postsurgical period. A two separates 10 cm VAS with 'no pain' at the left and 'unbearable pain' at the right end as verbal end points. Two forms for each day, one for the recipient site and one for the donor site. Forms were given to subjects after completion of the operation and they asked to mark the pain value they feel at the end of each day. Forms were collected on the day of suture removal (day 14).

The color matching between the graft and the adjacent tissue was determined and compared by using professional evaluation at the end of the final post-operative follow up visit (6 months). Two blinded examiners through Visual Analog Scale (VAS). Actually, VAS is a scale for measurement of subjective features, which are difficult to measure. The test and control areas were assessed for color matching of the grafted tissue with the adjacent keratinized gingiva between canines area. The results were esthetically graded in three groups of Poor [1-3], Moderate [4-6] and Good [7-9].

Patient's Satisfaction was measured by scale from 0 to 10 was filled by each patient where 0 is not satisfied, Little satisfied [1-3], Average satisfied [4-6] and highly satisfied [7-10] is fully satisfied by the outcome, this reading was recorded only at the end of the study 6 months post-surgically.

graft area measurement was performed with Java-based analyse programme (ImageJ, National Institutes of Health, Bethesda, Maryland, USA). For evaluation of the graft area, graft borders were drawn after inserting the known distance between two fixed points on periodontal probe (10 mm) by the number of pixels between these two points. All evaluations were repeated twice, and the average value of these two measurements was calculated at 1-, 3-, and 6- month follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* non-smoker,
* not taking any medication

Exclusion Criteria:

* Pregnant
* lactating women
* gingival pigmentation
* previous periodontal surgery

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-05 (Actual)

PRIMARY OUTCOMES:
visual analogue scale (VAS) pain score | 7 days
  visual analogue scale (VAS) pain score in donor and receipt sites
surface area and color match | 6 months
  Clinical photographs were used to measure the surface area of the graft in all follow up periods, and to assess the color matching between the grafted area and the adjacent tissue at the end of the final follow-up visit on 6-month period

CONTACTS AND LOCATIONS:
Locations (1):
- Jordan University of Science and Technology, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: Undecided